CLINICAL TRIAL: NCT05747378
Title: An In-depth Study Assessing Eczema Patients Experiences in Medical Trials
Brief Title: Finding Patterns In Clinical Trial Experiences of Patients With Eczema
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 82431237
Record Dates: First submitted 2023-02-17; First posted 2023-02-28 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-02

CONDITIONS: Eczema
Keywords: Eczema
MeSH Terms: conditions — Eczema

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Historically, participation in clinical trials has been skewed towards certain groups. However, research on the factors that influence participation, both positive and negative, is limited.

Eczema clinical trial patients help us identify these factors by sharing trial experiences during the course of the observational medical study.

This study will include a diverse group of participants to gather a wide range of information on clinical trial experiences. The collected data will then be used to benefit future eczema patients who are considering participating in a clinical study.

ELIGIBILITY:
Inclusion Criteria:

* Patient has been diagnosed with eczema
* Patient is 18 years old
* Patient has self-identified as planning to enroll in an observational clinical study

Exclusion Criteria:

* Patient does not understand, sign, and return consent form
* Patient is pregnant
* Inability to perform regular electronic reporting

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with eczema who are actively considering participating in a clinical trial, but have not yet completed enrollment and randomization.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Number of patients who decide to enroll in a clinical trial for eczema. | 3 months
Rate of patients who remain in an eczema clinical trial to completion. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Allen SJ, Jordan S, Storey M, Thornton CA, Gravenor MB, Garaiova I, Plummer SF, Wang D, Morgan G. Probiotics in the prevention of eczema: a randomised controlled trial. Arch Dis Child. 2014 Nov;99(11):1014-9. doi: 10.1136/archdischild-2013-305799. Epub 2014 Jun 19. PMID 24947281
- [Background] Sawangjit R, Dilokthornsakul P, Lloyd-Lavery A, Lai NM, Dellavalle R, Chaiyakunapruk N. Systemic treatments for eczema: a network meta-analysis. Cochrane Database Syst Rev. 2020 Sep 14;9(9):CD013206. doi: 10.1002/14651858.CD013206.pub2. PMID 32927498
- [Background] Spada F, Harrison IP, Barnes TM, Greive KA, Daniels D, Townley JP, Mostafa N, Fong AT, Tong PL, Shumack S. Recruitment of adults with moderate eczema for a randomised trial: Comparison of traditional versus modern methods. Australas J Dermatol. 2021 Nov;62(4):e510-e515. doi: 10.1111/ajd.13699. Epub 2021 Sep 3. PMID 34477217

DOCUMENTS (1):
  • Informed Consent Form (2023-02-17): https://cdn.clinicaltrials.gov/large-docs/78/NCT05747378/ICF_000.pdf